CLINICAL TRIAL: NCT03545061
Title: Dutch National Prospective EMR Cohort. Longterm Follow Up After EMR for Large Flat/Sessile Colonic Polyps, a Prospective Study.
Brief Title: Dutch National Prospective EMR Cohort
Acronym: DN-PEC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-4449
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Large Bowel Polyp

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Prospective Study: Longterm Follow Up until S2 (2nd surveillance) at 18 months after EMR for Large Flat/Sessile Colonic Polyps.

ELIGIBILITY:
Inclusion Criteria:

* Flat or sessile polyp morphology (Paris classification 0-IIa/b/c, Is)
* Polyp size >20 mm
* Therapy: EMR
* Age > 18 years old
* Written informed consent

Exclusion Criteria:

* Participation in a competing study, such as the "CLIPPER trial" (registration number: NL62949.091.17).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients with 1 or more large flat or sessile polyps of 2 cm or larger, located in the colon, that are removed with EMR. These will often be patients diagnosed in the scope of the National Colon Cancer Screening programme.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Complications | 30 days post EMR
  Delayed bleeding, perforation and postpolypectomy syndrome
Recurrence | 6 months (S1) and 18 months (S2) after EMR
  Pathological and endoscopical re-appearance of adenoma

CONTACTS AND LOCATIONS:
Overall Officials: E. Van Geenen, dr, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands